CLINICAL TRIAL: NCT02603341
Title: Pragmatic Randomized Trial of Proton vs. Photon Therapy for Patients With Non-Metastatic Breast Cancer: A Radiotherapy Comparative Effectiveness (RADCOMP) Consortium Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19115
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Photons; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photon (Active Comparator): Photon therapy: once a day, 5 days a week, for 5 to 7 weeks
  Interventions: Radiation: Photon
- Proton (Active Comparator): Proton therapy: once a day, 5 days a week, for 5 to 7 weeks
  Interventions: Radiation: Proton

INTERVENTIONS:
Radiation: Photon — Photon Therapy:once a day, 5 days a week, for 5 to 7 weeks
  Arms: Photon
Radiation: Proton — Proton Therapy: once a day, 5 days a week, for 5 to 7 weeks
  Arms: Proton

SUMMARY:
A pragmatic randomized clinical trial of patients with locally advanced breast cancer randomized to either proton or photon therapy and followed longitudinally for cardiovascular morbidity and mortality, health-related quality of life, and cancer control outcomes. Quality of life is the outcome measure for the estimated primary completion date of December, 2024, www.radcomp.org.

DETAILED DESCRIPTION:
Because no one knows which radiation treatment is best, if you decide to take part in this study, you will be randomly assigned to 1 of 2 treatment groups, and then you will begin radiation treatment according to usual medical practice. Randomly assigning you to a group helps makes sure that each group has a similar mix of patients and makes the study better - and is only done when doctors are not sure whether one treatment is better than the other. You have an equal chance of getting into either treatment group, like a coin flip. Both you and your doctor will be told which treatment you will get.

No matter which group patients are in, doctors will work very carefully to reduce the radiation to healthy tissues. Both groups will followed for at least 10 years after completing radiation therapy. The results of this study will help decide which radiation is best for future patients with your type of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females or males diagnosed with pathologically (histologically) proven invasive mammary carcinoma (ductal, lobular or other) of the breast who have undergone either mastectomy or lumpectomy with any type of axillary surgery or axillary sampling.
* For patients who have undergone lumpectomy, any type of mastectomy and any type of reconstruction (including no reconstruction) are allowed.
* For patients who have undergone lumpectomy, there are no breast size limitations.
* Patients with non-metastatic breast cancer are eligible. This includes American Joint Committee on Cancer (AJCC) 7th edition left- or right-sided breast cancer clinical or pathologic stage I, II, III or loco-regionally recurrent at time of diagnosis. For patients that receive neoadjuvant chemotherapy, AJCC 7th edition left- or right-sided breast cancer pathologic stage yp 0, I, II, III are eligible.
* Bilateral breast cancer is permitted. Patients with bilateral breast cancer will be stratified as left-sided.
* Must be proceeding with breast/chest wall and nodal radiation therapy including internal mammary node treatment.
* Must have a pertinent history/physical examination within 90 days prior to registration.
* Age ≥ 21 years
* ECOG Performance Status 0 - 2 (asymptomatic to symptomatic but capable of self-care) within 90 days prior to randomization.
* Confirmation that the patient's health insurance will pay for the treatment in this study (patients may still be responsible for some costs, such as co-pays and deductibles). If the patient's insurance will not cover a specific treatment in this study and the patient still wants to participate, confirmation that the patient would be responsible for paying for any treatment received.
* Patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 180 days prior to registration as documented in the medical record. HIV testing is not required for eligibility for this protocol.
* The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria

* Definitive clinical or radiologic evidence of metastatic disease, as documented by the treating institution.
* Prior radiotherapy to the ipsilateral chest wall or ipsilateral breast or thorax. Individuals with prior radiotherapy in the contralateral breast or chest wall are eligible.
* Any radiation therapy for the currently diagnosed breast cancer prior to randomization.
* Dermatomyositis with a CPK level above normal or with an active skin rash or scleroderma.
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1238 (Estimated)
Dates: Start 2016-04-06 (Actual); Primary Completion 2036-11 (Estimated); Study Completion 2036-11 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of proton therapy vs. photon therapy | 10 years
  Compare the effectiveness of proton vs. photon therapy in reducing major cardiovascular events (MCE), defined as atherosclerotic coronary heart disease or other heart disease death, myocardial infarction, coronary revascularization, or hospitalization for major cardiovascular event (heart failure, valvular disease, arrhythmia, or unstable angina).

SECONDARY OUTCOMES:
Disease Control | 5 years
  Compare the non-inferiority of proton vs. photon therapy in reducing ipsilateral breast cancer local-regional recurrence and in reducing any recurrence, defined as the first reported breast cancer recurrence of any type (local-regional or distant or cancer-specific mortality)
Patient-reported Body Image and Function, Fatigue and Other Measures of Health-related Quality of Life (HRQOL) | 5 years
  Compare the effectiveness of proton vs. photon therapy in improving patient-reported body image and function, fatigue and other measures of health-related quality of life (HRQOL) (anxiety, social roles, financial toxicity, general satisfaction) and adverse events.
Radiation Dose and Quality of Life and Cardiac Toxicity | 5 years
  Develop predictive models to examine the association of radiation dose distribution (to heart and other normal tissues) and major cardiovascular events and quality of life outcomes.
Long Term Survival | 15 years
  To assess longer-term rates of breast cancer specific and overall survival and development of second malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Bonnie Ky, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Shannon MacDonald, MD, Study Chair — Massachusetts General Hospital
Locations (40):
- United States (40):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - UC San Diego, San Diego, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami Sylvester Cancer Center at Coral Gables, Coral Gables, Florida
  - University of Miami Sylvester Cancer Center - Deerfield, Deerfield Beach, Florida
  - University of Florida Health, Gainesville, Florida
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Insititute, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Medicine Proton Center, Chicago, Illinois
  - Willis Knighton, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - McLaren Proton Therapy, Flint, Michigan
  - William Beaumont, Royal Oak, Michigan
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - RWJ University Hospital Hamilton, Hamilton, New Jersey
  - Cancer Institute of NJ, New Brunswick, New Jersey
  - ProCure Proton Therapy Center, Somerset, New Jersey
  - New York Proton Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals, Case Medical Center, Cleveland, Ohio
  - University Pointe, University of Cincinnati, West Chester, Ohio
  - Oklahoma University - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Pinnacle Health Cancer Institute, Harrisburg, Pennsylvania
  - Abramson Cancer Center at Penn Medicine, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Thompson Proton Center, Knoxville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Center for Proton Therapy, Irving, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Bekelman JE, Lu H, Pugh S, Baker K, Berg CD, Berrington de Gonzalez A, Braunstein LZ, Bosch W, Chauhan C, Ellenberg S, Fang LC, Freedman GM, Hahn EA, Haffty BG, Khan AJ, Jimenez RB, Kesslering C, Ky B, Lee C, Lu HM, Mishra MV, Mullins CD, Mutter RW, Nagda S, Pankuch M, Powell SN, Prior FW, Schupak K, Taghian AG, Wilkinson JB, MacDonald SM, Cahlon O; RadComp (Radiotherapy Comparative Effectiveness Consortium). Pragmatic randomised clinical trial of proton versus photon therapy for patients with non-metastatic breast cancer: the Radiotherapy Comparative Effectiveness (RadComp) Consortium trial protocol. BMJ Open. 2019 Oct 15;9(10):e025556. doi: 10.1136/bmjopen-2018-025556. PMID 31619413
- See also: Study website — http://www.radcomp.org